CLINICAL TRIAL: NCT04712370
Title: Comparison of Conventional Caudal Block, Ultrasound Guided Caudal Block and Ultrasound Guided Erector Spinae Block for Pediatric Hip Surgery
Brief Title: Conventional Caudal Block, Ultrasound Guided Caudal Block and Ultrasound Guided Erector Spinae Block for Pediatric Hip Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Eman Hamdy Abu-Shanab, Principal Investigator and Assistant lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 33143/05/19
Record Dates: First submitted 2021-01-11; First posted 2021-01-15 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Conventional Caudal Block; Ultrasound Guided Caudal Block; Ultrasound Guided Erector Spinae Block; Pediatric Hip Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional caudal block (Active Comparator): Patients of this group will receive the conventional method (blind technique without ultrasound) of caudal block
  Interventions: Procedure: Conventional caudal block
- Ultrasound-guided caudal block (Experimental): Patients of this group will receive caudal block using ultrasound.
  Interventions: Procedure: Ultrasound-guided caudal block
- Ultrasound guided erector spinae plane Block (Experimental): Patients of this group will receive ultrasound guided erector spinae plane Block at the level of the transverse process of the second lumbar vertebrae(L2) .
  Interventions: Procedure: Ultrasound guided erector spinae plane Block

INTERVENTIONS:
Procedure: Conventional caudal block — Patients of this group will receive (0.5ml/kg) (plain bupivacaine 0.25% injected in the caudal epidural space) by the conventional method (blind technique without ultrasound).
  Arms: Conventional caudal block
Procedure: Ultrasound-guided caudal block — Using ultrasound, patients of this group will receive (0.5ml/kg) (plain bupivacaine 0.25% injected in the caudal epidural space).
  Arms: Ultrasound-guided caudal block
Procedure: Ultrasound guided erector spinae plane Block — Under ultrasound guidance, patients of this group will receive (0.5ml/kg) (plain bupivacaine 0.25% injected beneath the erector spinae muscle sheath) at the level of the transverse process of the second lumbar vertebrae(L2).
  Arms: Ultrasound guided erector spinae plane Block

SUMMARY:
This study will be conducted to compare the efficacy and safety of ultrasound guided erector spinae block , ultrasound guided caudal block and conventional caudal block for pain management after pediatric hip surgery.

ELIGIBILITY:
Inclusion Criteria:

* Both sex
* ASA physical activity I, II
* Age 4-12 years
* Admitted for elective hip surgery.

Exclusion Criteria:

* Parents refusal
* Children with severe systemic disease
* ASA III or IV
* Children with previous neurological or spinal anomaly, coagulation disorders
* History of premature birth
* Infection at the block injection site
* History of allergy to local anesthetics
* Bilateral hip surgery.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Estimated)
Dates: Start 2021-01-16 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-10 (Estimated)

PRIMARY OUTCOMES:
Degree of pain intensity | First 24 hours postoperative
  To evaluate the pain scores by (FLACC) scale. (FLACC) scale will be assessed after surgery over 24 hours where (0 = Relaxed and comfortable, 1-3 = Mild discomfort, 4-6 = Moderate pain ,7-10 = Severe discomfort /pain)

SECONDARY OUTCOMES:
Changes in mean arterial blood pressure | Intraoperative and first 24 hours postoperative
  Mean arterial blood pressure will be recorded before block performance at T0, intraoperatively at 15 and 30 minutes, then every 30 min till the end of surgery and after surgery at T (0, 2, 4, 6, 12, 24 h).
Changes in heart rate | Intraoperative and first 24 hours postoperative
  Heart rate will be recorded before block performance at T0, intraoperatively at 15 and 30 minutes, then every 30 min till the end of surgery and after surgery at T (0, 2, 4, 6, 12, 24 h).
Amount of Analgesic required in the first day after surgery | First 24 hours postoperative
  The total dose of intravenous (IV) acetaminophen 15 mg/kg if FLACC scores between 2 and 4 at the first 24 h after surgery, and total dose of tramadol 1 mg/kg (IV) in case of FLACC score > 4.
Time to first rescue analgesic demand after surgery. | First 24 hours postoperative
  measured from the end of surgery till patient require analgesia.
Success rate of block | Intraoperative duration
  a successful block is defined as absence of significant changes in heart rate following surgical induction. Heart rate increase is not>20% of the basal levels. If the increase is>20%, the block is accepted as unsuccessful.
Duration of performing the block | Intraoperative duration
  Block performing time is defined as the period between the insertion of the needle and termination of local anesthetic administration
Incidence of complications | Intraoperative and first 24 hours postoperative
  Hypotension, bradycardia, postoperative nausea, vomiting, urinary retention, prolonged motor block, pruritus and local anesthetic systemic toxicity (LAST).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: For 1 year after the end of the study
Access Criteria: The principal investigator will review requests